CLINICAL TRIAL: NCT03210584
Title: Multimodal Evaluation of Cartilage Lesions of Patellofemoral Joint
Acronym: MULTICART
Status: Completed | Type: Observational
Sponsor: University Hospital, Grenoble (Other)
Collaborators: Clinical Investigation Centre for Innovative Technology Network (Network)
Responsible Party: Sponsor
Other Study IDs: 38 RC16.213
Record Dates: First submitted 2017-06-06; First posted 2017-07-07 (Actual); Last update posted 2018-09-11 (Actual); Status verified 2018-09

CONDITIONS: Knee Osteoarthritis
Keywords: Knee joint; Cartilage degeneration; Ultrasound imaging; Full-Field Optical Coherence Tomography; 9,4 Tesla MRI; Multimodal evaluation
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: None Retained — cartilage samples undergoing total knee arthroplasty procedure
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Imaging measurements: All subject of the study have a knee osteoarthritis (OA) and are going to have a knee prosthetic surgery with cartilage excision. Multimodal evaluation is conducted on ex vivo human cartilage samples (2 samples per patient are selected : healthy and severely degraded).

SUMMARY:
Evaluation and comparison of histological analysis, 9,4 tesla MRI, Full-Field Optical Coherence Tomography (FFOCT) and ultrasound-based navigation system for cartilage degeneration analysis of patellofemoral joint.

DETAILED DESCRIPTION:
Knee osteoarthritis (OA) is a common and debilitating chronic degenerative disease of the articular cartilage. Despite recent progress in the field of cartilage imaging, no routinely used clinical imaging modality has the ability to evaluate and monitor changes in cartilage degeneration. This observationnal, pilot, prospective, non randomized, uncontrolled, monocentric study aim to compare three of the most innovative imaging systems, namely the 9,4 Tesla MRI, the FFOCT (Full-Field Optical Coherence Tomography) and the ultrasound-based navigation system in order to image healthly to severely degraded human cartilage samples. All methods will be cross-correlated and compared with histological data considered as the gold standard.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years of age
* Knee prosthetic surgery indication with cartilage excision.

Exclusion Criteria:

* Subjects who refuse to sign a non-objection form

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with knee arthroplasty indication for medial femoro-tibial osteoarthristis at University Hospital, Grenoble
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2017-01 (Actual); Study Completion 2018-09 (Actual)

PRIMARY OUTCOMES:
Evaluation and comparison of histologic analysis, 9,4 Tesla MRI, FFOCT and ultrasound-based navigation system for cartilage lesions analysis of patellofemoral joint. | 6 months
  Correlation between Osteoarthritis Research Society International (OARSI) grades performed for different modalities

SECONDARY OUTCOMES:
Evaluation of 9,4 Tesla MRI reconstructions in early osteoarthritis evaluation using visual qualitative information parameter obtained from the Average Pathlength Maps (APM). | 6 months
  Correlation between MRI quantitative parameters and gold standard OARSI grade
Evaluation of FFOCT reconstructions in early osteoarthritis evaluation using visual qualitative information parameter. | 6 months
  Correlation between quantitative parameters from FFOCT and gold standard OARSI grade
Evaluation of navigation ultrasound in early osteoarthritis evaluation using visual qualitative information parameter. | 6 months
  Correlation between quantitative parameters from navigation ultrasound and gold standard OARSI grade
Evaluation of of 9,4 Tesla MRI reconstruction in early osteoarthritis evaluation using visual quantitative information parameter obtained for the Average Pathlength Maps. | 6 months
  Correlation between quantitative parameters from the Average Pathlength Maps and gold standard OARSI grade
Evaluation of FFOCT reconstructions in early osteoarthritis evaluation using visual quantitative information parameter. | 6 months
  Thickness average of cartilage
Evaluation of FFOCT reconstructions in early osteoarthritis evaluation using visual quantitative information parameter. | 6 months
  Roughness average of cartilage
Evaluation of navigation ultrasound in early osteoarthritis evaluation using visual quantitative information parameter. | 6 months
  Thickness average of cartilage
Inter-observer robustness analysis of the OARSI classification | 6 months
  Inter-observers Kappa coefficient
Intra-observer robustness analysis of the OARSI classification | 6 months
  Intra-observers Kappa coefficient

CONTACTS AND LOCATIONS:
Overall Officials: Alexandre Moreau-Gaudry, MD, PhD, Principal Investigator — Clinical Investigation Centre for Innovative Technology Network
Locations (1):
- Orthopedic Surgery Department, University Grenoble Hospital, Grenoble, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Clinical Investigation Centre for Innovative Technology Network website — http://www.cic-it.fr/cic-it-grenoble.php